CLINICAL TRIAL: NCT05915936
Title: Comparative Study of Laparoscopic Ventral Mesh Rectopexy Versus Perineal Stapler Resection for External Full-Thickness Rectal Prolapse in Elderly Patients: Enhanced Outcomes and Reduced Recurrence Rates - A Retrospective Cohort Study
Brief Title: LVMR Versus PSR for External FTRPin Elderly Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Tamer.A.A.M.Habeeb, professour of general and laparoscopic surgery, Zagazig University
Other Study IDs: rectal prolapse
Record Dates: First submitted 2023-06-07; First posted 2023-06-23 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Rectal Prolapse
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic ventral mesh rectopexy: correction of rectal prolapse through laparoscopic ventral mesh rectopexy
  Interventions: Procedure: LVMR
- perineal stapler resection: correction of rectal prolapse through perineal stapler resection
  Interventions: Procedure: PSR

INTERVENTIONS:
Procedure: LVMR — laoparoscopic ventral mesh rectopexy
  Groups: laparoscopic ventral mesh rectopexy
Procedure: PSR — perineal stapler resection
  Groups: perineal stapler resection

SUMMARY:
In frail patients with external full-thickness rectal prolapse (FTRP), the exact postoperative recurrence and functional result outcomes difference between Laparoscopic ventral mesh rectopexy (LVMR) and perineal stapler resection (PSR) have not been investigated, leading to ineffective treatment.

Objectives: Evaluating the efficacy of PSR versus LVMR for treating external FTRP in the elderly.

Design: This was a retrospective study that involved multiple centers. Settings: This study was conducted in the colorectal surgical units of our Universities' Hospitals Patients: 330 elderly patients divided into LVMR group (250), and PSR (80) between April 2012 and April 2019. Before and after surgery, patients were evaluated using the Wexner Incontinence Scale, the Altomare Constipation Scale, and the patient's satisfaction.

Main outcomes measurement: The primary outcome was the recurrence rate and risk factors of FTRP. Secondary outcomes were postoperative incontinence and constipation and patients' satisfaction.

DETAILED DESCRIPTION:
From March 2012 to March 2019, 330 frail Patients were evaluated retrospectively using a prospectively collected database in the colorectal surgical divisions of our universities' hospitals. Eligible patients were complete external FTRP (grade 5 according to Oxford prolapse) only or with ODS or FI secondary to FTRP, ≥ 60 years, both sex, ASA-Score I-III, and completed at least four-years follow-up. Exclusion criteria were < 60 years, incomplete medical records, concurrent colorectal procedures, multi-compartmental prolapse requiring combined operations, open abdominal rectopexy, megacolon, pregnancy, inflammatory bowel disease, unfit for general anesthesia, recurrent rectal prolapse, prior anal surgery, patients under systemic steroid therapy, connective tissue disease, abnormal thyroid function, prior pelvic surgery, diverticulosis/stricture of the colon, previous colorectal resectional surgery, neurological disease, connective tissue disorders, psychiatric disorders, Chronic opioid use.

Outcome Definitions and Measurements:

The primary outcome focused on RP incidence and risk factors. Secondary outcomes included postoperative FI, ODS, and patient satisfaction. Recurrence entailed the presence of recurrent FTRP during follow-up, determined by physical examination and additional imaging. Continence status relied on the Jorge-Wexner grading scale , encompassing five items with a total score ranging from 0(complete continence) to 20 (complete incontinence). To assess ODS, the Altomare score uses 8 Likert scales for a maximum of 31 points for severe constipation []. Postoperative morbidity was assessed by Clavien and Dindo classification []. The measurement of external FTRP was obtained by assessing the distance between the distal margin of the rectum and the anal margin during straining. Anal stenosis was defined as the narrowing of the orifice, characterized by the inability of a 12-mm colonoscopy or the passage of one finger through the constricted opening. [].

ELIGIBILITY:
Inclusion Criteria:

* complete external FTRP (grade 5 according to Oxford prolapse) only or with ODS or FI secondary to FTRP,
* ≥ 60 years,
* both sex,
* ASA-Score I-III, and
* completed at least four-years follow-up

Exclusion Criteria:

* < 60 years,
* incomplete medical records,
* concurrent colorectal procedures,
* multi-compartmental prolapse requiring combined operations,
* open abdominal rectopexy

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: elderly patients with complete FTRP
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2012-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
recurrent rate of rectal prolapse | 4 years
  % of recurrence after surgery

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Habeeb TAAM, Podda M, Chiaretti M, Kechagias A, Lledo JB, Kalmoush AE, Mustafa FM, Nassar MS, Labib MF, Teama SRA, Elshafey MH, Elbelkasi H, Alsaad MIA, Sallam AM, Ashour H, Mansour MI, Mostafa A, Elshahidy TM, Yehia AM, Rushdy T, Ramadan A, Hamed AEM, Yassin MA, Metwalli AM. Comparative study of laparoscopic ventral mesh rectopexy versus perineal stapler resection for external full-thickness rectal prolapse in elderly patients: enhanced outcomes and reduced recurrence rates-a retrospective cohort study. Tech Coloproctol. 2024 Apr 15;28(1):48. doi: 10.1007/s10151-024-02919-1. PMID 38619626